CLINICAL TRIAL: NCT02914665
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Cardiac and Renal Effects of Short Term Treatment With Elamipretide in Patients Hospitalized With Congestion Due to Heart Failure
Brief Title: A Phase 2 Study to Evaluate the Cardiac and Renal Effects of Short Term Treatment With Elamipretide in Patients Hospitalized With Congestion Due to Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIHF-204; 2016-000126-19 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-26 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
Keywords: Heart failure; diuresis; dropsy; congestion; elamipretide; MTP-131; Bendavia™
MeSH Terms: conditions — Heart Failure; Edema | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 mg elamipretide (Experimental): 20 mg elamipretide once daily for 7 consecutive days
  Interventions: Drug: elamipretide
- Placebo (Placebo Comparator): Placebo once daily for 7 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: elamipretide — 20 mg elamipretide administered intravenously once daily for 7 consecutive days
  Other Names: MTP-131, Bendavia
  Arms: 20 mg elamipretide
Drug: Placebo — Placebo administered intravenously once daily for 7 consecutive days
  Arms: Placebo

SUMMARY:
This is a phase 2 randomized, double-blind, placebo-controlled study to evaluate the cardiac and renal effects of short term treatment with elamipretide in patients hospitalized with congestion due to heart failure

ELIGIBILITY:
Inclusion Criteria:

* A history of chronic heart failure for at least 1 month
* Treated with ≥40 mg/day of furosemide or bumetanide ≥1 mg/day or torasemide ≥10 mg/day for at least 1 month
* In-hospital observation/admission and treatment for ≤72 hours and primary cause for admission is heart failure with persistent congestion in the opinion of the Investigator (i.e. at least +2 pitting oedema and/or an estimated 8 kg gain in weight over baseline over the past 4 weeks) requiring intravenous loop diuretic therapy
* Sufficiently severe oedema to justify treatment by an intravenous infusion of furosemide of 10 mg/hour for at least 48 hours
* Systolic blood pressure >90 mmHg and considered to be haemodynamically stable, in the opinion of the Investigator
* History of left ventricular ejection fraction (LVEF) ≤40% confirmed in the last 18 months
* NT-proBNP >1500 pg/ml or BNP >500 pg/ml
* An eGFR of >30 mL/min/1.73 m2 using the eGFR (mL/min/1.73 m2) = 175 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.212 if African American)

Exclusion Criteria:

* Acute coronary syndrome, stroke, or transient ischemic attack (TIA), coronary or peripheral revascularization procedures, valve procedures, OR any major surgical procedure within the previous 6 weeks
* Invasive cardiac investigation and/or treatment (i.e. coronary angiography, percutaneous coronary intervention [PCI] or surgery) or other surgical procedure planned in the next 4 weeks
* Use of intravenous radiographic contrast agent within 72 hours prior to screening or planned use during the study
* Severe, in the investigators opinion, uncorrected valve disease or congenital heart disease as the cause for cardiac decompensation
* Acute mechanical cause of decompensated heart failure such as papillary muscle rupture
* Obstructive or infiltrative cardiomyopathy (e.g. amyloid, sarcoid, etc), suspected acute myocarditis, or heart failure related to an untreated metabolic condition (e.g. haemochromatosis)
* Second or third degree heart block unless the subject has a ventricular pacemaker
* Atrial fibrillation/flutter with sustained ventricular response of >130 bpm
* Placement of a ventricular resynchronization device within the previous 6 weeks
* Treatment or planned treatment with intravenous inotropic agents other than digoxin at any time on this admission
* Receipt of intravenous vasodilator therapy ≤ 6 hours prior to randomization
* The presence of any mechanical assist device or listed for or a history of a heart transplant
* Severe respiratory disease or anticipated need for mechanical respiratory support (i.e. mechanical ventilation)
* Anuric in the previous 24 hours
* Haemoglobin <9 g/dL at screening or planned blood transfusions in the next 30 days
* Serum potassium >5.5 mEq/L
* Marked proteinuria suggestive of nephrotic syndrome
* Estimated GFR (eGFR) as per MDRD equation <30 ml/min
* Serum albumin of < 2.8 g/dL
* Liver enzymes (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) elevation >5 times the upper limit of normal (ULN)
* Total bilirubin >2.0 times ULN in the absence of Gilbert's Syndrome
* Current or planned ultrafiltration, paracentesis, haemofiltration or dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Change in NT-proBNP between Baseline and Day 8/Early Discharge | Baseline to Day 8

SECONDARY OUTCOMES:
Number of patients staying in the same functional renal function class measured with MDRD formula compared to the number of patients with decreasing or increasing renal function measured with MDRD formula | Baseline to Day 3 and Day 8
Number of patients showing a decrease in body weight compared to baseline as well as number of patients showing either no decrease or an increase in body weight compared to baseline | Baseline to Day 3 and Day 8
Calculation of decrease or increase in body weight normalised to the average dose (in mg) of furosemide administered | Baseline to Day 3 and Day 8
The patient and physician global assessment is a 7-point scale which either the patient or the physician will assess from 0 to 10 and will be mathematically averaged on a daily basis in order to compare the different averages throughout the study. | Baseline to Day 3 and Day 8
The average daily dose of diuretic (furosemide - adjusted for thiazide dose if administered) between baseline and Day 3 and Day 8/Early Discharge | Baseline to Day 3 and Day 8
All adverse events, serious adverse events and SUSARs will be summarised per treatment group, namely elamipretide versus placebo, and compared at the end of the study. | Baseline to Day 8
Half-life (T1/2) | Baseline to Day 8
Area under the concentration - time curve from 0-24 h (AUC 0-24) | Baseline to Day 8
Area under the concentration - time curve from 0- infinity (AUC 0-∞) | Baseline to Day 8
Peak Plasma Concentration (Cmax) | Baseline to Day 8

CONTACTS AND LOCATIONS:
Locations (46):
- Belgium (2):
  - Hospital Onze Lieve Vrouw campus Aalst, Aalst
  - Hospital ZNA Middelheim, Antwerp
- Bulgaria (6):
  - Department of Internal Diseases, "Multiprofile Hospital for Active Treatment Sveta Ekaterina - Dimitrovgrad" EOOD, Dimitrovgrad
  - Clinic of Cardiology, "Second Multiprofile Hospital for Active Treatement - Sofia" EAD, Sofia
  - Clinic of Cardiology, Multiprofile Hospital for Active Treatment National Heart Hospital" EAD, Sofia
  - Clinic of Cardiology, "City Clinic University Multiprofile Hospital for Active Treatment" EOOD, Sofia
  - Clinic of Internal Diseases, "Multiprofile Hospital for Active Treatment, "Sveta Anna Sofia" AD, Sofia
  - Department of Cardiology, "Multiprofile Regional Hospital for Active Treatement Dr. Stefan Cherkezov" AD, Veliko Tarnovo
- France (2):
  - Hôpital Henri Mondor, Créteil
  - CHU de Rangueil, Toulouse
- Hungary (4):
  - Hungarian Institute Of Cardiology, Department of Adult Cardiology, Budapest
  - Semmelweis University Heart and Vascular Center, Budapest
  - County St. George University Teaching Hospital, Department of Internal Medicine Cardiology, Székesfehérvár
  - Zala County Hospital Cardiology Department, Zalaegerszeg
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Riga East Clinical University Hospital, Clinic Gailezers, Liepāja
  - Liepaja Regional Hospital, Liepāja
  - Pauls Stradins Clinical University Hospital, Latvian Centre of Cardiology, Riga
- Netherlands (7):
  - Hospital Jeroen Bosch, 's-Hertogenbosch
  - Deventer Hospital, Deventer
  - Hospital Gelderse Vallei, Ede
  - University Medical Center Groningen, Groningen
  - Hospital Antonius/D&A research Genetic, Sneek
  - Hospital Elisabeth -Tweesteden, Tilburg
  - Hospitals Gelre, Zutphen
- Poland (3):
  - Bieganski Provincial Specialist Hospital, Department of Cardiology, Clinic of Cardiology UM, Lodz
  - Cardinal Stefan Wyszynski, Institute of Cardiology, Clinic Heart Failure and Transplantation, Warsaw
  - Cardinal Stefan Wyszynski, Institute of Cardiology, Clinic of Coronary Heart Disease and Structural Heart Disease, Warsaw
- Serbia (6):
  - Clinical Centre of Serbia, Emergency Centre, Belgrade
  - Clinical Centre of Serbia, Institute for Cardiovascular Diseases, Belgrade
  - Clinical Hospital Centre Bezanijska kosa, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Institute for Cardiovascular Diseases of Vojvodina, Kamenitz
  - Clinical Centre Nis, Niš
- Spain (9):
  - Complexo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Alvaro Cunqueiro, Pontevedra
  - Hospital Clínico Universitario de Valencia, Valencia
  - Consorci Hospital General Universitari de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (3):
  - Bradford Royal Infirmary, Bradford
  - Glenfield Hospital, Leicester
  - Torbay Hospital, Torquay